CLINICAL TRIAL: NCT05946135
Title: A Randomized, Double-blind, Active Controlled Clinical Trial to Evaluate the Efficacy of Fexuprazan for the Prevention or Control of Gastritis Symptoms in Patients on Treatment With Systemic Steroids (FEAST)
Brief Title: Efficacy of Fexuprazan for Prevention or Control of Gastritis Symptoms in Patients on Treatment With Systemic Steroids
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4-2023-0598
Record Dates: First submitted 2023-07-06; First posted 2023-07-14 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Patients on Treatment With Systemic Steroids
MeSH Terms: interventions — Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): lansoprazole + placebo for Fexuprazan Hydrochloride
  Interventions: Drug: Lansoprazole
- Intervention (Experimental): placebo for lansoprazole + Fexuprazan Hydrochloride
  Interventions: Drug: Fexuprazan Hydrochloride

INTERVENTIONS:
Drug: Lansoprazole — taking lansoprazole + placebo for Fexuprazan Hydrochloride for 4 weeks
  Arms: Control
Drug: Fexuprazan Hydrochloride — taking placebo for lansoprazole + Fexuprazan Hydrochloride for 4 weeks
  Arms: Intervention

SUMMARY:
* This clinical trial is conducted as a double-blind, randomized, and active drug control clinical trial. If the screening results determine that the selection/exclusion criteria are met, the clinical trial drugs are randomly assigned at a 1:1 ratio of the Pexuprazan 40 mg and the Lansoprazole 15 mg dose group and taken for 4 weeks.
* Gastritis symptoms are evaluated four weeks after baseline (Visit1) and clinical drug administration (Visit2), and if it is determined that gastritis is necessary according to the medical team's judgment due to gastrointestinal symptoms during the study participation period, endoscopy is performed to check whether gastritis occurs.

ELIGIBILITY:
Inclusion Criteria:

1. A person who voluntarily signed a consent form
2. Adult men and women over 20 years of age
3. Patients who require systemic steroid treatment of at least 4 weeks of moderate dose (20 mg/day or more based on prednisolone) due to respiratory diseases during screening

   * Patients who are already on steroids can also participate (If there is a gastric protective agent in use, patients should agree to replace it with clinical trial drug)
4. Patients who satisfy both of the following in relation to the evaluation index of gastritis symptoms during screening

   - Gastritis symptom frequency indicator: 5 points or less

   - Gastritis symptom intensity indicator: 5 points or less
5. A person who has at least one of the following risk factors for gastric ulcer during screening

   ① Long-term use of NSAIDs for longer than 12 weeks (NSAIDs should be maintained continuously during the clinical trial.)

   ② A person who has a history of peptic ulcer in the past

   ③ 50 years of age or older

   ④ In combination with low-dose aspirin (aspirin 325 mg/day or less) (Low-dose aspirin should be maintained continuously during the clinical trial.)
6. A person who understand and follow the guidance of the research manager according to the research plan, and who can participate whole period of clinical trial

Exclusion Criteria:

1. A person who has a hypersensitivity reaction to the components of this clinical trial drug or benzimidazole-based drug or has a history of clinically significant hypersensitivity reaction
2. A person who has undergone surgery that may affect gastric acid secretion, such as upper gastrointestinal resection, gastric acid secretion inhibition surgery, and gastric mucosal resection
3. Those who have a history of gastrointestinal malignancies within 5 years of screening (excluding after endoscopic resection of gastric carcinoma or early gastric cancer)
4. Patients with Barrett's esophagus (over 3 cm), gastroesophageal varices, esophageal stenosis, ulcer stenosis, active peptic ulcers, and acute gastrointestinal bleeding
5. Patients with inflammatory bowel disease (Crohn's disease, ulcerative colitis, etc.), irritable bowel syndrome (IBS), primary esophageal motility disorder, and pancreatitis
6. Patients with eosinophilic esophagitis (if the esophageal biopsy determines that it is not eosinophilic esophagitis, they can participate)
7. Those who have a history of gastric acid secretion disorders such as Zolinger-Elison syndrome
8. A person who is currently confirmed positive for Helicobacter pyrroly infection
9. Persons taking medications contraindicated to clinical trial drug (e.g., atazanavir, nelfinavir, or rilpivirine-containing agents)
10. Patients with genetic problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose absorption disorder
11. Patients with severe renal and liver disorders according to the physician's judgment
12. A person who disagrees with the appropriate use of contraception by himself/herself or his/her partner during the clinical trial period
13. Pregnant women or breast feeding women
14. Any person who has any clinical findings that are deemed medically inappropriate for this trial under the judgment of the research manager

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-11-07 (Actual); Primary Completion 2025-09-08 (Actual); Study Completion 2025-09-08 (Actual)

PRIMARY OUTCOMES:
Changes in baseline gastritis symptoms based on gastritis symptom index at 4 weeks | baseline and 4 weeks later
  To evaluate the effect of preventing gastritis symptoms, changes in gastritis symptoms using gastritis symptom index after 4 weeks compared to baseline were compared. The gastritic symptoms index consisted of 10 items to be questioned about the frequency and degree of symptoms over the past 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Ji Ye Jung, Principal Investigator — Severance Hospital, Division of Pulmonary and Critical Care Medicine
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No